CLINICAL TRIAL: NCT01214642
Title: A Phase 1 Dose-Escalation Study of LY2523355 in Patients With Advanced Cancer
Brief Title: A Dose-Escalation Study for Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11619; I1Y-MC-JFBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Cancer
MeSH Terms: conditions — Neoplasms | interventions — pegfilgrastim; litronesib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2523355 Days 1, 5, 9 (Experimental): LY2523355 administered intravenously on Days 1, 5 and 9, starting dose is 2 milligrams per meter squared (mg/m^2) for 2 planned 21-day cycles. Participants may continue on study drug until disease progression, unacceptable toxicity or other withdrawal criterion are met.
  Interventions: Drug: LY2523355
- LY2523355 Days 1, 8 (Experimental): LY2523355 administered intravenously on Days 1 and 8, starting dose is 8 mg/m^2 for 2 planned 21-day cycles. Participants may continue on study drug until disease progression, unacceptable toxicity or other withdrawal criterion are met.
  Interventions: Drug: LY2523355
- LY2523355 Days 1, 5 + pegfilgrastim (Experimental): LY2523355 administered intravenously on Days 1 and 5, starting dose is 8 mg/m^2 for 2 planned 21-day cycles and 6 mg pegfilgrastim administered subcutaneously on Day 6 of each 21-day cycle for the 2 planned cycles and for any subsequent cycles of LY2523355 received. Participants may continue on study drug until disease progression, unacceptable toxicity or other withdrawal criterion are met.
  Interventions: Drug: pegfilgrastim; Drug: LY2523355
- LY2523355 Days 1, 4 + pegfilgrastim (Experimental): LY2523355 administered on Days 1 and 4, starting dose is 12 mg/m^2 for 2 planned 21-day cycles and 6 mg pegfilgrastim administered subcutaneously on Day 5 of each 21-day cycle for the 2 planned cycles and for any subsequent cycles of LY2523355 received. Participants may continue on study drug until disease progression, unacceptable toxicity or other withdrawal criterion are met.
  Interventions: Drug: pegfilgrastim; Drug: LY2523355

INTERVENTIONS:
Drug: pegfilgrastim — Administered subcutaneously
  Arms: LY2523355 Days 1, 4 + pegfilgrastim; LY2523355 Days 1, 5 + pegfilgrastim
Drug: LY2523355 — Administered intravenously

SUMMARY:
This study is being conducted to determine the safety of LY2523355 for the treatment of advanced and/or metastatic cancer (including Non-Hodgkin's lymphoma).

DETAILED DESCRIPTION:
This study is a multi-center, non-randomized, open label, dose-escalation, Phase 1 study of intravenous LY2523355 in patients with advanced and/or metastatic cancer (including non-Hodgkin's lymphoma) for whom no treatment of higher priority exists.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of advanced and/or metastatic cancer (solid tumors or Non-Hodgkin's lymphoma) that is refractory to standard therapy or for which no proven effective therapy exists. Participants entering the dose confirmation phase (Part B) of the study must also have a tumor that is safely amenable to serial biopsies
* Have the presence of measurable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) or Revised International Working Group Lymphoma Response Criteria
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy, or other investigational therapy for at least 28 days (6 weeks for mitomycin-C or nitrosoureas) prior to study enrollment
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug
* Females with child bearing potential must have had a negative urine or serum pregnancy test less than or equal to 7 days prior to the first dose of study drug
* Have an estimated life expectancy of greater than or equal to 12 weeks.

Exclusion Criteria:

* Have symptomatic, untreated or uncontrolled central nervous system (CNS) metastases. Participants with treated CNS metastases are eligible provided their disease is radiographically stable, asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants. Screening of asymptomatic participants without history of CNS metastases is not required
* Have current acute or chronic leukemia
* Have had an autologous or allogenic bone marrow transplant
* Females who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A is the LY2523355 dose escalation phase and Part B is the LY2523355 dose confirmation phase. The reasons for discontinuation listed in the participant flow are the reasons the participant discontinued treatment and a participant was considered to have "completed" the trial if they received at 2 cycles of treatment.
Groups:
- Part A - Days 1, 5, 9 - 2 mg/m^2/Day: 2 milligrams per meter squared per day (mg/m^2/day) LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 5, 9 - 4 mg/m^2/Day: 4 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 5, 9 - 8 mg/m^2/Day: 8 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 5, 9 - 7 mg/m^2/Day: 7 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 5, 9 - 6 mg/m^2/Day: 6 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 5, 9 - 5 mg/m^2/Day: 5 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 8 - 8 mg/m^2/Day: 8 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 8 of 21-day cycle.
- Part A - Days 1, 5+PEG - 8 mg/m^2/Day: 8 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus pegfilgrastim (PEG) administered subcutaneously on Day 6.
- Part A and B- Days 1, 5+PEG - 12 mg/m^2/Day: 12 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6.
- Part A - Days 1, 5+PEG - 16 mg/m^2/Day: 16 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6.
- Part A - Days 1, 5+PEG - 14 mg/m^2/Day: 14 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6.
- Part B - Days 1, 4+PEG - 12 mg/m^2/Day: 12 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 4 of 21-day cycle plus PEG administered subcutaneously on Day 5.
Period: Overall Study
Arm/Group | Part A - Days 1, 5, 9 - 2 mg/m^2/Day | Part A - Days 1, 5, 9 - 4 mg/m^2/Day | Part A - Days 1, 5, 9 - 8 mg/m^2/Day | Part A - Days 1, 5, 9 - 7 mg/m^2/Day | Part A - Days 1, 5, 9 - 6 mg/m^2/Day | Part A - Days 1, 5, 9 - 5 mg/m^2/Day | Part A - Days 1, 8 - 8 mg/m^2/Day | Part A - Days 1, 5+PEG - 8 mg/m^2/Day | Part A and B- Days 1, 5+PEG - 12 mg/m^2/Day | Part A - Days 1, 5+PEG - 16 mg/m^2/Day | Part A - Days 1, 5+PEG - 14 mg/m^2/Day | Part B - Days 1, 4+PEG - 12 mg/m^2/Day
Started | 3 | 3 | 6 | 6 | 6 | 3 | 6 | 3 | 13 (All participants who received 12 mg/m2/day on Days 1 and 5 plus PEG in Part A and Part B.) | 4 | 4 | 6
Received at Least 1 Dose of Study Drug | 3 | 3 | 6 | 6 | 6 | 3 | 6 | 3 | 13 | 4 | 4 | 6
Complete at Least 2 Cycles of Study Drug | 3 | 1 | 5 | 4 | 6 | 1 | 6 | 3 | 12 | 2 | 2 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 6 | 6 | 6 | 3 | 6 | 3 | 13 | 4 | 4 | 6
Not completed — Progressive Disease | 3 | 2 | 3 | 5 | 5 | 3 | 5 | 3 | 10 | 2 | 1 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of LY2523355.
Groups:
- Part A and B - Days 1, 5+PEG - 12 mg/m^2/Day: 12 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6 in Part A and Part B.
- Total: Total of all reporting groups
Arm/Group | Part A - Days 1, 5, 9 - 2 mg/m^2/Day | Part A - Days 1, 5, 9 - 4 mg/m^2/Day | Part A - Days 1, 5, 9 - 8 mg/m^2/Day | Part A - Days 1, 5, 9 - 7 mg/m^2/Day | Part A - Days 1, 5, 9 - 6 mg/m^2/Day | Part A - Days 1, 5, 9 - 5 mg/m^2/Day | Part A - Days 1, 8 - 8 mg/m^2/Day | Part A - Days 1, 5+PEG - 8 mg/m^2/Day | Part A and B - Days 1, 5+PEG - 12 mg/m^2/Day | Part A - Days 1, 5+PEG - 16 mg/m^2/Day | Part A - Days 1, 5+PEG - 14 mg/m^2/Day | Part B - Days 1, 4+PEG - 12 mg/m^2/Day | Total
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 3 | 6 | 3 | 13 | 4 | 4 | 6 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.60 (5.484) | 48.07 (19.657) | 59.73 (7.541) | 61.67 (9.352) | 58.45 (12.425) | 56.73 (7.267) | 59.77 (6.959) | 67.10 (1.212) | 62.02 (7.598) | 57.10 (25.069) | 60.18 (10.205) | 59.43 (18.595) | 60.08 (11.471)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 1 | 4 | 3 | 2 | 2 | 4 | 2 | 3 | 2 | 30
  Male | 1 | 2 | 2 | 5 | 2 | 0 | 4 | 1 | 9 | 2 | 1 | 4 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 1 | 4 | 6 | 4 | 3 | 6 | 3 | 10 | 4 | 3 | 6 | 51
  African | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
  Hispanic | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6
  East Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  West Asian (Indian sub-continent) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 6 | 6 | 3 | 6 | 3 | 13 | 4 | 4 | 6 | 63

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose and Schedule for Phase 2 Studies
Description: The recommended dose and schedule for Phase 2 studies is defined as the maximum tolerated dose (MTD). MTD is defined as the dose level at which no more than 2 dose limiting toxicities (DLTs), no more than 3 dose reductions (DR) or dose omissions (DO) and no more than 1 DLT plus 2 DR/DO occurred. DLT is defined as an adverse event (AE) occurring in Cycle 1 with the following criteria according to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0: Any ≥Grade 3 nonhematological toxicity (except nausea/vomiting or diarrhea controlled with treatment or fatigue); ≥Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia with bleeding; Grade 4 hematological toxicity of >5 days duration, excluding thrombocytopenia; febrile neutropenia.
Time Frame: Cycle 1 (21 days): Day 1, 5 and 9, any AE reported
Population: All participants who received at least 1 dose of LY2523355.
Measure: Number; unit: mg/m^2/day
Groups:
- LY2523355 / LY2523355 +PEG: Escalating doses starting at 2 milligrams per meter squared per day (mg/m^2/day) LY2523355 administered by intravenous infusion over 1 hour on Days 1, 5, and 9; escalating doses starting at 8 mg/m^2/day LY2523355 administered by intravenous infusion over 1 hour on Days 1 and 8 or Days 1 and 5 plus 6 mg pegfilgrastim (PEG) administered subcutaneously on Day 6; or 12 mg/m^2/day LY2523355 administered by intravenous infusion over 1 hour on Days 1 and 4 plus 6 mg PEG administered subcutaneously on Day 5 of 21-day cycle for 2 planned cycles and any subsequent cycle up to 38 cycles of 21-days. The maximum allowed dose was 30 mg/m^2/day.
Arm/Group | LY2523355 / LY2523355 +PEG
Number analyzed (Participants) | 63
mg/m^2/day | 8

2. Secondary Outcome: Number of Participants With Clinically Significant Effects
Description: Clinically significant effects were defined as serious and other non-serious adverse events (AEs). A summary of serious and other non-serious AEs is located in the Reported Adverse Events module.
Time Frame: Baseline to Cycle 38 (21-day cycles): daily for AEs
Population: All participants who had at least 1 dose of LY2523355.
Measure: Count of Participants; unit: Participants
Groups:
- Part A - Days 1, 5+PEG - 8 mg/m2/Day: 8 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus pegfilgrastim (PEG) administered subcutaneously on Day 6.
- Part A - Days 1, 5+PEG - 12 mg/m^2/Day; Part B - Days 1, 5+PEG - 12 mg/m^2/Day: 12 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6.
- Part B - Days 1, 4+PEG - 12 mg/m^2/d: 12 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 4 of 21-day cycle plus PEG administered subcutaneously on Day 5.
Arm/Group | Part A - Days 1, 5, 9 - 2 mg/m^2/Day | Part A - Days 1, 5, 9 - 4 mg/m^2/Day | Part A - Days 1, 5, 9 - 8 mg/m^2/Day | Part A - Days 1, 5, 9 - 7 mg/m^2/Day | Part A - Days 1, 5, 9 - 6 mg/m^2/Day | Part A - Days 1, 5, 9 - 5 mg/m^2/Day | Part A - Days 1, 8 - 8 mg/m^2/Day | Part A - Days 1, 5+PEG - 8 mg/m2/Day | Part A - Days 1, 5+PEG - 12 mg/m^2/Day | Part A - Days 1, 5+PEG - 16 mg/m^2/Day | Part A - Days 1, 5+PEG - 14 mg/m^2/Day | Part B - Days 1, 5+PEG - 12 mg/m^2/Day | Part B - Days 1, 4+PEG - 12 mg/m^2/d
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 3 | 6 | 3 | 3 | 4 | 4 | 10 | 6
Participants
  Serious AEs | 1 | 2 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 4 | 4
  Other Non-Serious AEs | 3 | 2 | 6 | 6 | 6 | 3 | 6 | 3 | 3 | 4 | 4 | 10 | 6

3. Secondary Outcome: Pharmacokinetics Maximum Concentration (Cmax), Single Dose
Description: Plasma Cmax following a single dose of LY2523355 at each dose level across all schedules and in the presence or absence of pegfilgrastim (PEG).
Time Frame: Cycle 1 Day 1 of 21-day cycle: Predose, 1 hour (hr), 2,4,6,8,24,48 and 72 hr postdose
Population: All participants who received 1 dose of LY2523355 and had Cmax samples collected on Day 1 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- 2 mg/m^2/Day LY2523355: 2 milligrams per meter squared per day (mg/m^2/day) LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- 4 mg/m^2/Day LY2523355: 4 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- 5 mg/m^2/Day LY2523355: 5 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- 6 mg/m^2/Day LY2523355: 6 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- 7 mg/m^2/Day LY2523355: 7 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- 8 mg/m^2/Day LY2523355: 8 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion across all schedules and in the presence or absence of PEG administered subcutaneously.
- 12 mg/m^2/Day LY2523355: 12 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6 and on Days 1 and 4 of 21-day cycle plus PEG administered subcutaneously on Day 5.
- 14 mg/m^2/Day LY2523355: 14 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6.
- 16 mg/m^2/Day LY2523355: 16 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6.
Arm/Group | 2 mg/m^2/Day LY2523355 | 4 mg/m^2/Day LY2523355 | 5 mg/m^2/Day LY2523355 | 6 mg/m^2/Day LY2523355 | 7 mg/m^2/Day LY2523355 | 8 mg/m^2/Day LY2523355 | 12 mg/m^2/Day LY2523355 | 14 mg/m^2/Day LY2523355 | 16 mg/m^2/Day LY2523355
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 15 | 19 | 4 | 4
nanograms/milliliter (ng/mL) | 45.2 (25) | 126 (31) | 137 (81) | 196 (40) | 218 (26) | 192 (32) | 379 (10) | 598 (32) | 463 (43)

4. Secondary Outcome: Pharmacokinetics Maximum Concentration (Cmax), Multiple Dose
Description: Plasma Cmax following multiple doses of LY2523355 at each dose level across all schedules and in the presence or absence of pegfilgrastim (PEG).
Time Frame: Cycle 1 Days 4, 5, 8 or 9 of 21-day cycle:Predose, 1 hour (hr), 2,4,6,8,24,48 and 72 hr postdose
Population: All participants who received 2 doses of study drug and had a Cmax sample collected on Days 4, 5, 8 or 9 of Cycle 1 (based on schedule of administration) after multiple dose administration of LY2523355.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | 2 mg/m^2/Day LY2523355 | 4 mg/m^2/Day LY2523355 | 5 mg/m^2/Day LY2523355 | 6 mg/m^2/Day LY2523355 | 7 mg/m^2/Day LY2523355 | 8 mg/m^2/Day LY2523355 | 12 mg/m^2/Day LY2523355 | 14 mg/m^2/Day LY2523355 | 16 mg/m^2/Day LY2523355
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 4 | 11 | 19 | 4 | 4
nanograms/milliliter (ng/mL) | 49.1 (15) | 121 (58) | 196 (43) | 124 (40) | 200 (69) | 186 (42) | 367 (35) | 415 (46) | 485 (45)

5. Secondary Outcome: Pharmacokinetics Area Under the Concentration-time Curve (AUC), Single Dose
Description: Plasma AUC from time zero to infinity [AUC(0-∞)] and AUC from time zero to 24 hours post-dose [AUC(0-24)] following a single dose of LY2523355 at each dose level across all schedules and in the presence or absence of pegfilgrastim (PEG).
Time Frame: Cycle 1 Days 4, 5, 8 or 9 of 21-day cycle:Predose, 1 hour (hr), 2,4,6,8,24,48 and 72 hr postdose
Population: All participants who received 1 dose of LY2523355 and had pharmacokinetic samples collected on Day 1 of Cycle 1 to enable calculation of AUC(0-∞) and AUC(0-24).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliter (ng*hr/mL)
Groups:
- 5 mg/m^2/Day LY25233552: 5 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
Arm/Group | 2 mg/m^2/Day LY2523355 | 4 mg/m^2/Day LY2523355 | 5 mg/m^2/Day LY25233552 | 6 mg/m^2/Day LY2523355 | 7 mg/m^2/Day LY2523355 | 8 mg/m^2/Day LY2523355 | 12 mg/m^2/Day LY2523355 | 14 mg/m^2/Day LY2523355 | 16 mg/m^2/Day LY2523355
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 15 | 19 | 4 | 4
nanograms*hour/milliter (ng*hr/mL)
  AUC(0-∞) | 158 (55) | 517 (71) | 584 (70) | 648 (45) | 758 (32) | 669 (28) | 1400 (41) | 2050 (23) | 1900 (28)
  AUC(0-24) | 106 (47) | 351 (63) | 366 (57) | 507 (30) | 566 (32) | 513 (27) | 1040 (37) | 1620 (24) | 1400 (26)

6. Secondary Outcome: Pharmacokinetic Areas Under the Concentration Time Curve (AUC), Multiple Dose
Description: Plasma AUC from time zero to infinity (0-∞) and AUC from time zero to 24 hours (0-24) post-dose following multiple doses of LY2523355 at each dose level across all schedules and in the presence or absence of pegfilgrastim (PEG).
Time Frame: Cycle 1 Days 4, 5, 8 or 9 of 21-day cycle:Predose, 1 hour (hr), 2,4,6,8,24,48 and 72 hr postdose
Population: All participants who received 2 doses of study drug and had pharmacokinetic samples collected on Day 4, 5, 8, or 9 of Cycle 1 (based on schedule of administration) to enable calculation of AUC(0-∞) and AUC(0-24) after multiple dose administration of LY2523355.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | 2 mg/m^2/Day LY2523355 | 4 mg/m^2/Day LY2523355 | 5 mg/m^2/Day LY2523355 | 6 mg/m^2/Day LY2523355 | 7 mg/m^2/Day LY2523355 | 8 mg/m^2/Day LY2523355 | 12 mg/m^2/Day LY2523355 | 14 mg/m^2/Day LY2523355 | 16 mg/m^2/Day LY2523355
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 4 | 11 | 19 | 4 | 4
nanograms*hour/milliliter (ng*hr/mL)
  AUC(0-∞) | 172 (34) | 377 (73) | 718 (52) | 356 (43) | 717 (66) | 575 (38) | 1340 (49) | 1280 (43) | 1510 (36)
  AUC(0-24) | 130 (27) | 308 (77) | 508 (34) | 298 (37) | 562 (66) | 452 (37) | 956 (40) | 1110 (46) | 1230 (26)

7. Secondary Outcome: Number of Participants With Tumor Response
Description: Response was assessed using Response Evaluation Criteria In Solid Tumors (RECIST) criteria and the Revised International Working Group (IWG) lymphoma response criteria for lymphoma patients. Complete Response (CR) was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions; Partial Response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD) was defined as at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase over nadir. Tumor response is CR + PR.
Time Frame: Baseline to measured disease progression or discontinuation up to Cycle 38 (21-day cycles)
Population: All participants who received 1 dose of LY2523355.
Measure: Number (90% Confidence Interval); unit: participants
Groups:
- LY2523355 Days 1, 5 and 9: Escalating dose started at 2 milligrams per meter squared (mg/m^2) LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5 and 9, for two planned cycles of 21 days. Dose could be escalated by a maximum increment of the lesser of doubling the current dose or 4 milligrams per meter squared per day (mg/m^2/day), with a maximum allowed dose of 30 mg/m^2/day. Participants continued on study drug until disease progression, unacceptable toxicity or other withdrawal criterion were met up to 38 cycles of 21 days.
- LY2523355 Days 1 and 8: Escalating dose started at 8 mg/m^2 of LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 8 for two planned 21-day cycles. Dose could be escalated by a maximum of 4 mg/m^2/day, with a maximum allowed dose of 30 mg/m^2/day. Participants continued on study drug until disease progression, unacceptable toxicity or other withdrawal criterion were met up to 38 cycles of 21-days.
- LY2523355 Days 1 and 5 + PEG: Escalating dose started at 8 mg/m^2 LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5, for two planned cycles of 21-days and 6 mg pegfilgrastim (PEG) administered subcutaneously on Day 6 of each 21-day cycle for the 2 planned cycles and for any subsequent cycles of LY2523355 received. Dose could be escalated by a maximum of 4 mg/m^2/day, with a maximum allowed dose of 30 mg/m^2/day. Participants continued on study drug until disease progression, unacceptable toxicity or other withdrawal criterion were met up to 38 cycles of 21-days.
- LY2523355 Days 1 and 4 + PEG: 12 mg/m^2 LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 4, for two planned 21 days cycles, 6 mg PEG administered subcutaneously on Day 5 of each 21-day cycle for the 2 planned cycles and for any subsequent cycles of LY2523355 received. Participants continued on study drug until disease progression, unacceptable toxicity or other withdrawal criterion were met up to 38 cycles of 21-days.
Arm/Group | LY2523355 Days 1, 5 and 9 | LY2523355 Days 1 and 8 | LY2523355 Days 1 and 5 + PEG | LY2523355 Days 1 and 4 + PEG
Number analyzed (Participants) | 27 | 6 | 24 | 6
participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Groups:
- Part A - Days 1, 5, 9 - 2 mg/m^2/Day: Part A (Dose Escalation Phase): 2 milligrams per meter squared per day (mg/m^2/day) LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 5, 9 - 4 mg/m^2/Day: Part A (Dose Escalation Phase): 4 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 5, 9 - 8 mg/m^2/Day: Part A (Dose Escalation Phase): 8 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 5, 9 - 7 mg/m^2/Day: Part A (Dose Escalation Phase): 7 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 5, 9 - 6 mg/m^2/Day: Part A (Dose Escalation Phase): 6 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 5, 9 - 5 mg/m^2/Day: Part A (Dose Escalation Phase): 5 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1, 5, and 9 of 21-day cycle.
- Part A - Days 1, 8 - 8 mg/m^2/Day: Part A (Dose Escalation Phase): 8 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 8 of 21-day cycle.
- Part A - Days 1, 5+PEG - 8 mg/m^2/Day: Part A (Dose Escalation Phase): 8 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus pegfilgrastim (PEG) administered subcutaneously on Day 6.
- Part A - Days 1, 5+PEG - 12 mg/m^2/Day: Part A (Dose Escalation Phase): 12 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6.
- Part A - Days 1, 5+PEG - 16 mg/m^2/Day: Part A (Dose Escalation Phase): 16 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6.
- Part A - Days 1, 5+PEG - 14 mg/m^2/Day: Part A (Dose Escalation Phase): 14 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6.
- Part B - Days 1, 5+PEG - 12 mg/m^2/Day: Part B (Dose Maintenance Phase): 12 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 5 of 21-day cycle plus PEG administered subcutaneously on Day 6.
- Part B - Days 1, 4+PEG - 12 mg/m^2/d: Part B (Dose Maintenance Phase): 12 mg/m^2/day LY2523355 administered intravenously as a 1-hour infusion on Days 1 and 4 of 21-day cycle plus PEG administered subcutaneously Day 5.
Arm/Group | Part A - Days 1, 5, 9 - 2 mg/m^2/Day | Part A - Days 1, 5, 9 - 4 mg/m^2/Day | Part A - Days 1, 5, 9 - 8 mg/m^2/Day | Part A - Days 1, 5, 9 - 7 mg/m^2/Day | Part A - Days 1, 5, 9 - 6 mg/m^2/Day | Part A - Days 1, 5, 9 - 5 mg/m^2/Day | Part A - Days 1, 8 - 8 mg/m^2/Day | Part A - Days 1, 5+PEG - 8 mg/m^2/Day | Part A - Days 1, 5+PEG - 12 mg/m^2/Day | Part A - Days 1, 5+PEG - 16 mg/m^2/Day | Part A - Days 1, 5+PEG - 14 mg/m^2/Day | Part B - Days 1, 5+PEG - 12 mg/m^2/Day | Part B - Days 1, 4+PEG - 12 mg/m^2/d
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 2/6 | 2/6 | 1/6 | 0/3 | 1/6 | 0/3 | 0/3 | 3/4 | 2/4 | 4/10 | 4/6
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 6/6 | 6/6 | 6/6 | 3/3 | 6/6 | 3/3 | 3/3 | 4/4 | 4/4 | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Days 1, 5, 9 - 2 mg/m^2/Day (N=3) | Part A - Days 1, 5, 9 - 4 mg/m^2/Day (N=3) | Part A - Days 1, 5, 9 - 8 mg/m^2/Day (N=6) | Part A - Days 1, 5, 9 - 7 mg/m^2/Day (N=6) | Part A - Days 1, 5, 9 - 6 mg/m^2/Day (N=6) | Part A - Days 1, 5, 9 - 5 mg/m^2/Day (N=3) | Part A - Days 1, 8 - 8 mg/m^2/Day (N=6) | Part A - Days 1, 5+PEG - 8 mg/m^2/Day (N=3) | Part A - Days 1, 5+PEG - 12 mg/m^2/Day (N=3) | Part A - Days 1, 5+PEG - 16 mg/m^2/Day (N=4) | Part A - Days 1, 5+PEG - 14 mg/m^2/Day (N=4) | Part B - Days 1, 5+PEG - 12 mg/m^2/Day (N=10) | Part B - Days 1, 4+PEG - 12 mg/m^2/d (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A - Days 1, 5, 9 - 2 mg/m^2/Day (N=3) | Part A - Days 1, 5, 9 - 4 mg/m^2/Day (N=3) | Part A - Days 1, 5, 9 - 8 mg/m^2/Day (N=6) | Part A - Days 1, 5, 9 - 7 mg/m^2/Day (N=6) | Part A - Days 1, 5, 9 - 6 mg/m^2/Day (N=6) | Part A - Days 1, 5, 9 - 5 mg/m^2/Day (N=3) | Part A - Days 1, 8 - 8 mg/m^2/Day (N=6) | Part A - Days 1, 5+PEG - 8 mg/m^2/Day (N=3) | Part A - Days 1, 5+PEG - 12 mg/m^2/Day (N=3) | Part A - Days 1, 5+PEG - 16 mg/m^2/Day (N=4) | Part A - Days 1, 5+PEG - 14 mg/m^2/Day (N=4) | Part B - Days 1, 5+PEG - 12 mg/m^2/Day (N=10) | Part B - Days 1, 4+PEG - 12 mg/m^2/d (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 5 (5) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 3 (3) | 5 (5) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 7 (7) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Central line infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cortisol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calcium ionised decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prothrombin time ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep talking (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penile oedema (Reproductive system and breast disorders) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/5 (0) | 0/2 (0) | 0/0 (0) | 1/4 (1) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 0/7 (0) | 0/4 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/5 (0) | 0/2 (0) | 0/0 (0) | 1/4 (1) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 0/7 (0) | 0/4 (0)
Testicular swelling (Reproductive system and breast disorders) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/5 (0) | 0/2 (0) | 0/0 (0) | 0/4 (0) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 1/7 (1) | 0/4 (0)
Vulval disorder (Reproductive system and breast disorders) | 0/2 (0) | 0/1 (0) | 0/4 (0) | 0/1 (0) | 1/4 (1) | 0 (0) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 0/2 (0) | 0/3 (0) | 0/3 (0) | 0/2 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/2 (0) | 0/1 (0) | 1/4 (1) | 0/1 (0) | 0/4 (0) | 0 (0) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 0/2 (0) | 0/3 (0) | 0/3 (0) | 0/2 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days